CLINICAL TRIAL: NCT00861627
Title: Phase 2 Study of Intravenous Administration of Reovirus Serotype 3 - Dearing Strain (REOLYSIN®) in Combination With Paclitaxel and Carboplatin in Patients With Metastatic or Recurrent Non-Small Cell Lung Cancer Who Have KRAS or EGFR Activated Tumors
Brief Title: Phase 2 Study of REOLYSIN® in Combination With Paclitaxel and Carboplatin for Non-Small Cell Lung Cancer With KRAS or EGFR Activation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 016
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Non-small Cell Lung
Keywords: REOLYSIN; reovirus; non-small cell lung cancer; carcinoma; oncolytics virus; chemotherapy; paclitaxel; carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — reolysin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: REOLYSIN® — 3x10E10 TCID50, 1 hour intravenous infusion, administered on Days 1, 2, 3, 4 and 5 of a 21 day cycle
  Other Names: reovirus serotype 3 Dearing Strain
Drug: Carboplatin — 5 AUC mg/mL min, 30 min intravenous infusion, given on Day 1 of a 21 day cycle
Drug: Paclitaxel — 175 mg/m2, 3 hour intravenous infusion, given on Day 1 of 21 day cycle

SUMMARY:
The purpose of this Phase 2 study is to investigate whether intravenous administration of a wild type reovirus (REOLYSIN®) in combination with paclitaxel and carboplatin is effective and safe in the treatment of Non-Small Cell Lung Cancer with KRAS or EGFR activation.

DETAILED DESCRIPTION:
Reovirus Serotype 3 - Dearing Strain (REOLYSIN®) is a naturally occurring, ubiquitous, non-enveloped human reovirus. Reovirus has been shown to replicate selectively in Ras-transformed cells causing cell lysis. Activating mutations in ras or mutation in oncogenes signaling through the ras pathway may occur in as many as 80% of human tumors. The specificity of the reovirus for Ras-transformed cells, coupled with its relatively nonpathogenic nature in humans, makes it an attractive anti-cancer therapy candidate.

Given the ability of reovirus to replicate and cause oncolysis in Ras-activated cells, the high incidence of K-ras mutations in lung cancers, and the Ras-mediated activation often encountered in EGFR-addicted tumors, the administration of REOLYSIN® in combination with chemotherapy is expected to result in enhanced clinical benefit in non-small cell lung cancer (NSCLC) patients with K-ras mutations and/or EGFR aberrant activation in their tumors. Patients with de novo or acquired EGFR mutations in their tumors that confer resistance to EGFR TKIs (e.g. T790) are expected to benefit as well. This is a single arm, open-label, Phase 2 study of REOLYSIN® given intravenously with paclitaxel and carboplatin every 3 weeks (21 days is defined as a cycle) in NSCLC patients with tumors driven by these pathways.

Paclitaxel at a dose of 175 mg/m2 will be given i.v. as a 3 hour infusion on Day 1 followed by carboplatin given i.v. AUC 5 mg/mL•minute. REOLYSIN® will be given over 60 min on Day 1 (starting after completion of the carboplatin infusion), and on Days 2 - 5. The treatment cycle will be repeated every 21 days.

Patients will receive 4 to 6 cycles of paclitaxel and carboplatin, at the treating physician's discretion according to standard of practice, in conjunction with REOLYSIN®. After completion of the 4 to 6 cycles of paclitaxel and carboplatin, REOLYSIN® may be continued as monotherapy Days 1-5 of each 21 day cycle until there is evidence of disease progression or unacceptable toxicity. Patients may continue to receive therapy under this protocol, provided they have not experienced either progressive disease or unacceptable drug-related toxicity that does not respond to either supportive care or dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* have histologically or cytologically confirmed stage IIIB (pleural effusion; IVA on revised IASLC staging) or stage IV, or recurrent, non-small cell lung cancer with evidence of RAS- or EGFR- activation in their tumors, as defined by EGFR activating mutations in exons 18 to 21, EGFR FISH amplification, or K-ras mutations in exon 2 (codons 12,13,61).
* have evidence of measurable disease. For patients previously irradiated, the measurable lesion(s) must be outside of the treated field.
* be chemotherapy naïve for their metastatic or recurrent NSCLC. Prior adjuvant chemotherapy or chemo-XRT for treatment of localized disease is allowed, provided it has been ≥ 6 months since the last chemotherapy infusion. Previous radiation for palliative purposes is also allowed, as long as it has been ≥4 weeks from the last dose.
* Patients who have been previously treated with EGFR tyrosine kinase inhibitors as their only systemic treatment are eligible, provided this treatment has been discontinued for ≥4 weeks. Patients who have received erlotinib as first line treatment without chemotherapy and experience tumor progression will be eligible.
* have NO continuing acute toxic effects (except alopecia) of any prior radiotherapy, chemotherapy, or surgical procedures, i.e., all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, version 3.0) Grade ≤ 1. Surgery (except biopsies) must have occurred at least 28 days prior to study enrollment.
* have an ECOG Performance Score of ≤ 2.
* have a life expectancy of at least 3 months.
* have baseline laboratory results as follows:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10E9 [SI units 10^9/L]
  * Platelets ≥ 100 x10E9 [SI units 10E9/L] (without platelet transfusion)
  * Hemoglobin ≥ 9.0 g/dL [SI units gm/L] (with or without RBC transfusion)
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Bilirubin ≤ 1.5 x ULN
  * AST/ALT ≤ 2.5 x ULN
  * Negative pregnancy test for females of childbearing potential.
* be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.

Exclusion Criteria:

* Receive concurrent therapy with any other anticancer agent while on study.
* Received chemotherapy within 6 months, or radiotherapy or EGFR therapy within 4 weeks, prior to entering the study or have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Have brain metastases. Patients with resected oligometastasis are eligible if post resection MRI demonstrates resolution. Gamma knife treated patients are also eligible, if there are no more than two treated metastases confined to the same area of the brain and a post treatment MRI shows a decrease in the metastases.
* Have ≥ grade 2 peripheral neuropathy at baseline.
* Have uncontrolled cardiac dysfunction, including a myocardial infarction in the preceding 6 months, or known cardiac ejection fraction < 40%.
* Be on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* Be a pregnant or breast-feeding woman. Female patients of childbearing potential must agree to use effective contraception, must be surgically sterile, or must be postmenopausal. Male patients must agree to use effective contraception or be surgically sterile. Barrier methods are a recommended form of contraception.
* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/ social situations that would limit compliance with study requirements.
* Have dementia or altered mental status that would prohibit informed consent.
* Have any other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-03; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Determine the objective response rate (complete response (CR) + partial response (PR)) of the treatment regimen in the study population | For PR or CR, changes in tumor measurements must be confirmed 4 weeks after the criteria for response are first met.

SECONDARY OUTCOMES:
Determine the median duration of progression-free survival of patients receiving the study treatment. | during and following study
Determine the median to 1-year survival of patients receiving the study treatment. | up to one year
Evaluate the safety and tolerability of REOLYSIN® in combination with paclitaxel and carboplatin in this patient population. | within 30 days of last dose of REOLYSIN®
Determine the proportion of patients receiving the above treatment who are alive and free of disease progression at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villalona, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - The Ohio State University Medical Center, James Cancer Hospital and Solove Research Institute, Columbus, Ohio